CLINICAL TRIAL: NCT04086004
Title: Additional Effects of Motor Imagery Practice With Dual Task Training in Stroke Patients
Brief Title: Dual Task Balance Training With Additional Motor Imagery Practice in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maria Zafar REC/00554
Record Dates: First submitted 2019-09-04; First posted 2019-09-11 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Stroke
Keywords: Motor Imagery practice; Stroke; Dual task training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I Experimental Motor Imagery (Experimental): Motor imagery practice
  Interventions: Other: Group I Experimental Motor Imagery
- Group II Dual Task Training (Experimental): Dual-task balance training
  Interventions: Other: Dual task training

INTERVENTIONS:
Other: Group I Experimental Motor Imagery — The experimental group will receive dual task balance training for 30 minutes/day with additional mental imagery for 10 minutes/day, three days/week, for a period of eight weeks
  Other Names: Group II Experimental Dual Task Training
  Arms: Group I Experimental Motor Imagery
Other: Dual task training — group will receive dual task balance training for 40 minutes for three days/ week for eight weeks
  Arms: Group II Dual Task Training

SUMMARY:
The importance of potent rehabilitation with dual task balance and gait training is improving and also there have been divergent opinions about the effectiveness of Motor Imagery on balance and gait function. Dual tasking has also proved beneficial results on stroke patients. Mental stimulation with task performance is a new intervention.. So the purpose of my study is to investigate the combination of Motor Imagery Practice and dual task rehabilitative training on balance and gait targeting the population of post stroke patients

DETAILED DESCRIPTION:
Stroke is a disease which occurs when the blood flow to the brain is cut off due to hemorrhage or ischemia in the blood vessels.Stroke is the second leading cause of death and a major cause of disability worldwide. Its incidence is increasing because the population ages . The quantity of individuals influenced by stroke will unavoidably ascend as global life expectancy increases. The frequency of motor deficits following a stroke can be up to 80% in a defined elderly population. Only a small percentage of this group (approximately 20%) will partially recover from impaired motor ability, leaving approximately 50-60% who are left with some form of chronic motor deficiency the burden of stroke seems to be high in Pakistan as in other south Asian countries. Not only the mean age of patients with stroke is less compared to patients in the developed world, approximately 20% of patients are under the age of 45 years. Hypertension is by far the most common risk factor also in young stroke patients. Hypertension and other conventional risk factors are highly prevalent in the country.To function in daily life, an individual must be able to maintain and adopt various postures, react to external disturbances, and use automatic postural responses that precede voluntary movements. A major focus of rehabilitation programs, therefore, is to improve balance and optimize function and mobility.Balance is the ability to maintain the body's center of mass over its base of support. Balance is a term used to describe the ability of a person to maintain or move within a weight-bearing posture without falling.Stroke patients experience various symptoms such as sensory disorder ,mobility defects and cognitive disorder which negatively affect functions for carrying out activities of daily living.The inability of stroke survivors to swing the involved leg rapidly might be the most critical factor adding to the enormous number of falls to the paretic side.balance and gait ability revival is a critical goal in stroke rehabilitation. A variety of interventions, such as virtual reality, robotics and mental practice with motor imagery, have been studied to improve the gait ability of stroke patients.Cognitive-motor and motor dual tasks assume significant role in day by day life: strolling while at the same time talking, utilizing a cell phone, carrying a pack or watching traffic.The dual-task program is effective in improving dual-task mobility, reducing falls and fall-related injuries in ambulatory chronic stroke patients with intact cognition. During dual-tasking, individuals with stroke have shown more pronounced performance decreasing in either the cognitive, mobility, or both tasks, compared with healthy older adults (ie, cognitive-motor interference) Mental practice is a new rehabilitation method that refers to the mental rehearsal of motor imagery content with the goal of improving motor performance.Motor imagery training is a helpful elective methodology for physical recovery following stroke, and offers protected, accessible, and cheap treatment strategy that is the utilization at home without specific equipments. Motor imagery training is free from physical execution of a disabled limb, and takes into account utilization of the mind to in restoring the circuitry that mediates voluntary movement. The preparation can make cortical plasticity changes like those made after physical action, in this way, these systems point to the capability of utilizing motor imagery practice in the neurological recovery of people following stroke.Hui yang cho et al concluded that Gait training with motor imagery training improves the balance and gait abilities of chronic stroke patients significantly better than gait training alone . According to recent study, conducted by Young Hyeon Bae et al. concluded that specific balance training with motor imagery is much beneficial and improve both balance and gait. Gye Yeop Kim et al found that dual-task training improves cognitive and walking abilities of patients with stroke.In another study conducted by Gui Bin Song et al reported that dual task training is more effective for increasing balance ability.

ELIGIBILITY:
Inclusion Criteria:

* Modified Rankin scale disability level 2-3
* Sub acute and chronic stroke patients.
* Ability to walk independently over ground for at least 10 m with or without use of an assistive device
* absence of any cognitive impairment
* No significant body or visual spatial hemi-neglect,
* Good ability for imagery functioning (a score of 32 or higher on the revision of Movement Imagery Questionnaire)

Exclusion Criteria:

-The patient will be excluded if he/she reported serious visual or somatosensory, orthopedic impairments.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | Change from Baseline balance to 8 Weeks
  The Berg balance scale (BBS) is used to assess the participant's ability to retain stability. The BBS is a widely used test for the assessment of elderly population with impairment of balance and individuals with neurological disorder while sitting, standing, and transferring. This test included both static and dynamic type task. The BBS uses a five-point ordinal scale ranging from 0 (disability) to 4(complete independent performance) and consists of 14 components; the maximum score is 56 points. The scale has been shown to be reliable and valid in stroke patients. A cut-off score of 45 points is used for fall prediction. The BBS involves 14 tasks; a total score of 56. Equipment required for this test were a stop watch or watch with a second's hand and a ruler or other indicator of 2, 5, and 10 inches. Excellent reliability (ICC range, 0.98-0.99) has been found in individuals with stroke survivors for BBS
Timed Up and Go test | Change from Baseline balance and mobility to 8 Weeks
  The Timed Up and Go (TUG) test was designed for the evaluation of balance and Measures mobility in people who are able to walk on their own (assistive device permitted) to find out the risk of fall . The subjects will be required to stand up from a chair, walk 3 m, turn around, return to the chair, and sit down. The time taken to complete this task will be measured. The test will be informed three times. The time required to complete this task will be measured from a stopwatch. The average values from 3 trials, with 1-min rest between each trial, were used for data analysis. This test has excellent reliability (ICC > 0.95) with stroke survivors
Functional reach Test: | Change from Baseline balance to 8 Weeks
  The patient is instructed to stand alongside a wall, however not contacting, a wall and position the arm that is nearer to the wall at 90 degrees of shoulder flexion with a closed fist. The assessor records the beginning position at the third metacarpal head on the measuring stick. Teach the patient to "Reach the extent that you can forward without taking a step." The area of the third metacarpal is recorded before and after a maximal forward reach. The mean score of three successful trials was calculated. Test-retest reliability of FR is high (interclass correlation coefficient (ICC) = 0.92) as interrater reliability is (ICC = 0.98)

SECONDARY OUTCOMES:
Fugl Meyer Scale (FMS) | Change from Baseline to 8 Weeks
  Changes from the Baseline this scale was measured
  Fugl Meyer Assessment is the utmost extensively used and approved clinical scale for assessment of sensorimotor loss in post stroke patients.This scale is comprised of five domains and there are 155 items in total:
  * Motor functioning (in the upper and lower extremities)
  * Sensory functioning (evaluates light touch on two surfaces of the arm and leg, and position sense for 8 joints)
  * Balance (contains 7 tests, 3 seated and 4 standing)
  * Joint range of motion (8 joints)
  * Joint pain 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
  MAS detecting the changes in muscle tone in patients with stroke.. It's a 6 point scale. 0=no muscle tone, 4= affected parts rigid flexion or extension.Its reliability is 0.567.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MsNMPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Railway General Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker C, Brouwer BJ, Culham EG. Use of visual feedback in retraining balance following acute stroke. Phys Ther. 2000 Sep;80(9):886-95. PMID 10960936
- [Background] Khealani BA, Hameed B, Mapari UU. Stroke in Pakistan. J Pak Med Assoc. 2008 Jul;58(7):400-3. PMID 18988415
- [Background] Kim SS, Lee HJ, You YY. Effects of ankle strengthening exercises combined with motor imagery training on the timed up and go test score and weight bearing ratio in stroke patients. J Phys Ther Sci. 2015 Jul;27(7):2303-5. doi: 10.1589/jpts.27.2303. Epub 2015 Jul 22. PMID 26311971
- [Background] Kenyon LK, Blackinton MT. Applying motor-control theory to physical therapy practice: a case report. Physiother Can. 2011 Summer;63(3):345-54. doi: 10.3138/ptc.2010-06. Epub 2011 Aug 10. PMID 22654241
- [Background] Melzer I, Goldring M, Melzer Y, Green E, Tzedek I. Voluntary stepping behavior under single- and dual-task conditions in chronic stroke survivors: A comparison between the involved and uninvolved legs. J Electromyogr Kinesiol. 2010 Dec;20(6):1082-7. doi: 10.1016/j.jelekin.2010.07.001. Epub 2010 Aug 2. PMID 20675152